CLINICAL TRIAL: NCT01511822
Title: Clinical, Metabolic and Endocrine Effects of the Treatment With Drospirenone and Ethinyl Estradiol Alone or in Combination With Myo-inositol in Young Women With Polycystic Ovary Syndrome (PCOS) and Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Dros_Myo2012
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: PCOS; Polycystic Ovary Syndrome
Keywords: PCOS; Insulin resistance; Hyperandrogenism; Myo-inositol
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Hyperandrogenism | interventions — drospirenone and ethinyl estradiol combination

ARMS (3):
- Drospirenone + Ethinyl estradiol (Active Comparator)
  Interventions: Drug: Drospirenone Ethinyl estradiol
- Drospirenone + Ethinyl estradiol + Myo-inositol (Experimental)
  Interventions: Drug: Drospirenone Ethinyl estradiol Myo-inositol
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Drospirenone Ethinyl estradiol — Drospirenone 3mg/die Ethinyl estradiol 30 mg/die (21 days/month for 6 months)
  Arms: Drospirenone + Ethinyl estradiol
Drug: Drospirenone Ethinyl estradiol Myo-inositol — Drospirenone 3mg/die Ethinyl estradiol 30 mg/die (21 days/months for 6 months) + Myo-inositol 6g /die for 6 months
  Arms: Drospirenone + Ethinyl estradiol + Myo-inositol
Drug: placebo
  Arms: Placebo

SUMMARY:
Polycystic ovary syndrome (PCOS) is a heterogeneous syndrome with a variety of metabolic and endocrine abnormalities and clinical symptoms.

The primary defect in PCOS consists of an abnormal androgen synthesis and secretion, particularly by ovarian theca cells. Insulin resistance and obesity may act as triggers, explaining the frequent association of PCOS with these metabolic conditions. Hyperinsulinaemia, which results from insulin resistance, stimulates both ovarian and adrenal androgen secretion and suppresses sex hormone-binding globulin synthesis from the liver. It results in an increase in free, biologically active androgens which are related to clinical signs such as hirsutism, acne, seborrhea, and alopecia.

Combined oral contraceptive (COC) therapy is a common treatment for PCOS and it was widely used in this group of patients providing clinical improvement in the areas of excessive hair growth, unpredictable menses, acne, and weight gain.

More recent studies outlined a deficiency in myo-inositol in women with PCOS and insulin-resistance. Myo-inositol is a precursor for many inositol-containing compounds and it plays critical and diverse roles in signal transduction, membrane biogenesis, vesicle trafficking, and chromatin remodeling. It is a precursor in the synthesis of phosphatidylinositol polyphosphates (PIPs) that are a source of several second messengers.

It has been reported that the administration of myo-inositol reduces serum insulin, decreases serum testosterone and enhances ovulation.

Due to the different beneficial actions, the aim of the present study is to evaluate the clinical, metabolic and endocrine effects of treatment with COC (drospirenone and ethinyl estradiol)alone or in combination with myo-inositol, in young women with PCOS and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Women fulfilled two out of three diagnostic criteria for PCOS, according to the 2003 Rotterdam Consensus conference
* Women with PCOS, insulin resistance, acne, hirsutism and seborrhea

Exclusion Criteria:

* Women with pre-existing secondary endocrine disorders
* Women wishing to conceive during the next 12 months
* Women with contradictions to oral contraceptive use
* Women with personal history of hypertension, diabetes mellitus or cardiovascular disorders
* Women who received treatment with oral contraceptives, or other drugs for the previous 6 months before entering the study.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult

PRIMARY OUTCOMES:
Score acne (acne grading system by Cook et al)
Score hirsutism (Ferriman-Gallwey classification)
Measurement of sex hormones in serum
Oral glucose tolerance test (OGTT)
Measurement of blood glucose and insulin levels
BMI

SECONDARY OUTCOMES:
Number of patients with adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto di Patologia Ostetrica e Ginecologica, Catania, Italy

REFERENCES:
- [Background] D'Anna R, Di Benedetto V, Rizzo P, Raffone E, Interdonato ML, Corrado F, Di Benedetto A. Myo-inositol may prevent gestational diabetes in PCOS women. Gynecol Endocrinol. 2012 Jun;28(6):440-2. doi: 10.3109/09513590.2011.633665. Epub 2011 Nov 28. PMID 22122627
- [Background] Minozzi M, Costantino D, Guaraldi C, Unfer V. The effect of a combination therapy with myo-inositol and a combined oral contraceptive pill versus a combined oral contraceptive pill alone on metabolic, endocrine, and clinical parameters in polycystic ovary syndrome. Gynecol Endocrinol. 2011 Nov;27(11):920-4. doi: 10.3109/09513590.2011.564685. Epub 2011 Mar 21. PMID 21417594
- [Background] Mathur R, Levin O, Azziz R. Use of ethinylestradiol/drospirenone combination in patients with the polycystic ovary syndrome. Ther Clin Risk Manag. 2008 Apr;4(2):487-92. doi: 10.2147/tcrm.s6864. PMID 18728832